CLINICAL TRIAL: NCT05206721
Title: The Effect of Suction System Flushing With Chlorhexidine on the Occurrence of Ventilator-Associated Pneumonia Among Mechanically Ventilated Patients
Brief Title: Open Suction Circuit Flushing With Chlorhexidine Decreases Ventilator-Associated Pneumonia: A Quasi-experimental Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Hesham Eid, Assistant Lecturer, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 245/2020
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Chlorhexidine; Endotracheal suctioning; Airway managment; suction circuit flushing
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Open tracheal suction system flushing with chlorhexidine
- Control group (No Intervention)

INTERVENTIONS:
Other: Open tracheal suction system flushing with chlorhexidine — After suctioning the patient's secretions, the responsible nurse inserted the SC into the CHX filled container and flushed the entire suction system with CHX.
  Arms: Intervention group

SUMMARY:
Background: Standard practice of flushing saline over the patient's secretions following suctioning is similar to pouring water over grease, leading to motivating bacterial colonization and proliferation inside the suctioning circuit (i.e., catheter, tube, and collecting jar), which can then migrate to patient's lung during suctioning procedure causing ventilator-associated pneumonia (VAP). Therefore, flushing this circuit using an appropriate disinfectant to prevent bacterial colonization inside it and thus decreasing pneumonia occurrence has been our crucial investigation idea.

Aim: To investigate the effect of suction system flushing with chlorhexidine (CHX) on the occurrence of VAP among mechanically ventilated patients (MVPs). Design: This study adopted a quasi-experimental research design, and a convenience sampling technique was used to recruit 136 patients to conduct this study. Setting: This study was conducted at surgical intensive care units of Mansoura University Emergency Hospital, Egypt. Results: The intervention group patients had a lower incidence of VAP (by 48.12%) compared with the control group. Moreover, the proposed technique was more effective in decreasing the incidence of late-VAP more than early-VAP. Furthermore, CHX reduced the cost of suction system flushing by 75%. Conclusion: Suction system flushing with CHX can significantly reduce the occurrence of VAP among MVPs and reduce the flushing cost. Therefore, this study recommends incorporating CHX into the daily care of MVPs.

DETAILED DESCRIPTION:
Research question Does OTSS flushing with CHX reduce the occurrence of VAP among MVPs?

Hypothesis OTSS flushing with CHX will reduce the occurrence of VAP among MVPs compared with traditional flushing using normal saline.

Aim This study aimed to investigate the effect of OTSS flushing with CHX on the occurrence of VAP among MVPs.

Research design A quasi-experimental research design was adopted to conduct this study. The subjects were randomly assigned to either the intervention or control group, and comparative results were analyzed based upon pre-post intervention follow-up for both groups.

Setting This study was conducted at the surgical ICUs affiliated with a university hospital in Egypt with 201-bed capacity. There are three surgical ICUs participated in the study; each one has 10 beds and provides care to patients with surgical and neurological problems, and multiple trauma injuries. These units are well equipped with advanced technology required for high quality patients' care. The nurse-patient ratio in these units is nearly 1:2.

Participants Patients admitted to the ICUs who were intubated within the previous 24 hours and were expected to receive MV support for more than 48 hours were recruited in the study. Excluded were patients diagnosed with pneumonia at the time of admission and/or having a Modified Clinical Pulmonary Infection Score (MCPIS) of 5 or greater, patients who had contraindications to suctioning (i.e., severe hemoptysis, increased intracranial pressure, and cerebrospinal fluid leaks), patients with pulmonary edema, acute respiratory distress syndrome (ARDS) and atelectasis because of their pulmonary infiltrate disease pathophysiology. Additionally, patients known to be allergic to CHX were also excluded.

Sample size calculation The sample size was calculated through DSS Research using a sample size calculator software, at 5% α error (95.0% significance) and 20.0% β error (80.0% power of the study). The sample size needed for the study was 136 patients and the patients were randomly assigned (the even number in the patients' list was assigned to the intervention group and the odd number to the control group) into two groups (68 in each group): The intervention group received CHX as the flushing solution for the OTSS. The control group received normal saline as the flushing using.

Instruments

Two tools were used to collect data for this study:

Tool Ι: "MVPs' assessment Tool"

This tool was developed by the primary investigator (PI) after reviewing relevant literature (14,17,18). The tool consists of three parts:

Part Ι: "Patients' Socio-demographic and health relevant Data" This part contained participants' sociodemographic data including age, gender, occupation, educational level, and smoking habits. Moreover, it covered the participants' health-relevant data, including the date and reason of ICU admission, medical diagnosis, past medical history, length of ICU stay, and modified Glasgow Coma Scale (GCS) score.

Part ΙΙ: "Ventilator modalities data" This part included the MV initiation date, artificial airway used, intubation process (e.g., urgent; or elective), endotracheal tube (ETT) size, and mode and duration of MV.

Part ΙΙΙ: "Endotracheal suctioning data" This part included the size of SC, type of SC connector, and duration of the total suctioning procedure.

Tool ΙΙ: "VAP diagnostic criteria sheet" This tool was adopted from Singh et al (19) and was used to assess the patients for clinical diagnosis of VAP. It included the MCPIS based on five clinical assessments; each variable is worth 0-2 points including the patient's body temperature, number of white blood cells, purulence and quantity of tracheal secretions (i.e., rare secretions, abundant, and purulent abundant secretions), oxygenation (calculated as PaO2 divided by the fraction of inspired oxygen "FiO2"), and chest radiography finding (i.e., no infiltrates, diffused infiltrates and localized infiltrates). The points for each variable of the MCPIS were summed, yielding a total score varied from 0 to 10 for data analysis.

Validity and reliability The content validity of tool I was assessed by seven experts from the Critical Care and Emergency Nursing and Medical fields. Accordingly, essential modifications were applied. Tool II was adopted and has been extensively used in many studies, which suggesting its validity. The overall reliability of the tool was tested using Cronbach's alpha test and was 0.798, indicating that the tool was reliable.

Pilot study A pilot study was conducted on 10% of the total sample (14 patients) before starting the data collection to evaluate the tools' clarity, feasibility, and applicability. Participants in the pilot study were excluded from the main study sample.

Data collection Official permission to conduct the study was obtained from the responsible authorities of the study setting after providing a detailed explanation of the study. The PI interviewed the patients' families on the first day of the patients' admission, during official ICU visiting hours, and explained to them the nature of the study. Once the next of kin agreed to allow the patient to participate in the study, the data collection process was commenced.

Procedure This study was conducted through three phases: assessment, implementation, and evaluation.

Assessment phase During this phase, an initial assessment was performed by the PI on the first day for all MVPs using MCPIS to confirm that they did not have pneumonia on admission, and they were free from the exclusion criteria using tool II "VAP diagnostic criteria sheet".

Implementation phase The PI did not develop a suctioning performance checklist according to standard guidelines or even ask the staff nurses to modify their current suctioning practices neither in the study group nor in the control group. This is to ensure that VAP occurrence was related to the use of CHX as the flushing solution for the suction system effect and not the modified suctioning technique.

A. Estimating the necessary CHX flushing amount The appropriate amount of CHX gluconate 0.2% solution required for effective OTSS flushing was investigated by the PI through clinical trials under the supervision of clinical expertise. The results showed that 40 mL CHX solution was an adequate amount for OTSS flushing and removal of any stacked secretions in the suction tube with a length of 1 m and catheter size of 16 Fr (Appendix I).

B. OTSS flushing intervention was performed through the following technique:

The intervention group:

Step I: Although allergic reactions to CHX are relatively rare, a sensitivity test was performed for the intervention group patients.

Step II: Routine suctioning technique (following the hospital's protocol) was performed on the patients by the responsible nursing staff.

Step III: The responsible nurse poured 40 mL CHX 0.2% solution from the CHX bottle into a sterile container (40 mL was marked by the second line in the container).

Step IV: After suctioning the patient's secretions, the responsible nurse inserted the SC into the 40 mL CHX filled container and flushed the entire suction system with CHX.

The control group:

Following the same above-mentioned steps II, III, and IV. Using traditional normal saline instead of CHX for OTSS flushing.

Evaluation phase MCPIS was calculated on the 3rd day for E-VAP and the 6th day for L-VAP. The minimum score was 0, and the maximum score was 10. Patients who obtained scores above 5 were diagnosed with pneumonia, and those who got scores below 5 were considered free of pneumonia.

For patients who obtained a score of 5 (borderline) with hemodynamic stability, the PI reevaluated them after 2 more days (8th day). Besides, for hemodynamically unstable patients, the PI ordered a sputum culture for them on the 6th day to verify their score. Patients with negative culture results obtained 0 points upon their score (MCPIS = 5) and were considered free of VAP, whereas those with positive results obtained 2 more points upon their score (MCPIS = 7) and were considered to have VAP.

Statistical analysis:

The obtained data were coded, computed, and statistically analyzed using Statistical Package for the Social Sciences (SPSS), version 24. Data were presented as frequency and percentages (qualitative variables) and mean ± standard deviation (quantitative continuous variables). Chi-square was used for comparing categorical variables and was replaced with Fisher's exact test (FET) or Monte Carlo exact test if the expected value of any cell was less than 5. Student's t-test was used for comparing continuous quantitative variables (two groups). For continuous quantitative variables that were not normally distributed, median was used as a central tendency measure. The Mann -Whitney U-test (Z) was used to compare the two groups. The difference was considered significant at P ≤ 0.05.

Ethical considerations Ethical approval was obtained from the Local Research Ethical Committee (Ref. No. 245/2020). Informed consent was obtained from the patients' families (next of kin), who were informed about the study, including the aim, procedure, benefits, and risks. The voluntariness nature of participation and the right to withdraw at any time without responsibility were also emphasized to them. Furthermore, the confidentiality of the participants' personal information was maintained.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the afore-mentioned ICUs who were intubated within the previous 24 hours and were expected to receive MV support for more than 48 hours were recruited in the study.

Exclusion Criteria:

* Patients with a clinical diagnosis of pneumonia at the time of admission and/or modified CPIS of 5 or greater.
* Patients who were previously intubated during the current hospital admission.
* Patients who had contraindications to suctioning such as severe hemoptysis, increased intracranial pressure, and cerebrospinal fluid leaks.
* Patients with pulmonary edema, ARDS, and those with atelectasis were also excluded from the study because of their pulmonary infiltrate disease pathophysiology.
* Patients known to be allergic to CHX were also eliminated from the study.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-11-19 (Actual)

PRIMARY OUTCOMES:
VAP Incidence | an average of 7 months
  Occurrence of Ventilator Associated Pneumonia

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Eid MH, Tantu MM, Latour JM, Sultan MA, Kandeel NA. Suction circuit flushing with chlorhexidine decreases ventilator-associated pneumonia: a quasi-experimental study. Front Med (Lausanne). 2023 Dec 4;10:1295277. doi: 10.3389/fmed.2023.1295277. eCollection 2023. PMID 38111699